CLINICAL TRIAL: NCT02248922
Title: An 8 Week Open-label Interventional Multicenter Study to Evaluate the Lung Clearance Index as Endpoint for Clinical Trials in Cystic Fibrosis Patients ≥ 6 Years of Age, Chronically Infected With Pseudomonas Aeruginosa
Brief Title: Evaluation of Lung Clearance Index in Cystic Fibrosis (CF) Patients, Infected With P.Aeruginosa
Acronym: ELIXIR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Reason for termination was challenge with enrollment and recruitment. A significant decrease in the eligible patient population was main driver.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTBM100CDE02
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-01

CONDITIONS: Chronic Lung Infection With Pseudomonas Aeruginosa in Cystic Fibrosis
Keywords: Cystic Fibrosis, Pseudomonas aeruginosa, Lung Clearance Index, Multiple Breath Washout, Inhaled Tobramycin, Inhaled Antibiotics.
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Lysine Acetyltransferase 5

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tobramycin ALL (Experimental): 300mg nebulized Tobramycin (Tobramycin inhalation solution(TIS)) or TOBI Podhaler (Tobramycin inhalation powder(TIP), equivalent dry powder)twice a day (BID) 28days on / 28 days off
  Interventions: Drug: TIS or TIP

INTERVENTIONS:
Drug: TIS or TIP — 300mg nebulized Tobramycin (Tobramycin inhalation solution(TIS)) or TOBI Podhaler (Tobramycin inhalation powder(TIP), equivalent dry powder)

SUMMARY:
The purpose of the study was to evaluate lung clearance index (LCI) by a standardized procedure in a well characterized study setting and to assess feasibility of LCI as a more sensitive method than forced expiratory volume at 1 second (FEV1) to measure effectiveness of antibiotic therapy in patients with CF aged 6 years and older with mild to moderate lung disease.

DETAILED DESCRIPTION:
This study was terminated prematurely. The reason for trial termination was challenge with enrollment and patient recruitment. A significant decrease in the eligible patient population had been identified as main driver.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF
* Patients with elevated LCI of ≥ 7.5 at screening
* Patients with FEV1 of ≥ 50% predicted at screening
* Use of inhaled Tobramycin in a 28 days on / off regimen in the past 3 months before screening
* chronic lung Infection with Pseudomonas aeruginosa

Exclusion Criteria:

* Patients who are regularly receiving more than one class of inhaled anti-pseudomonal antibiotic
* Patients who have used oral or intravenous anti-pseudomonal antibiotics within 28 days prior to on-phase of study drug
* Pregnant or nursing (lactating) women
* Change in dose, formulation or strength of the study drug in the past treatment cycle before screening
* History of hearing loss or chronic tinnitus
* Infection with Burkholderia cenocepacia complex

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Ziegler, PhD, Study Director — Novartis Pharma GmbH, Nürnberg, Germany
Locations (6):
- Germany (6):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Germering
  - Novartis Investigative Site, Jena

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Sutharsan S, Naehrig S, Mellies U, Sieder C, Ziegler J. An 8 week open-label interventional multicenter study to explore the lung clearance index as endpoint for clinical trials in cystic fibrosis patients >/=8 years of age, chronically infected with Pseudomonas aeruginosa. BMC Pulm Med. 2020 Jun 12;20(1):167. doi: 10.1186/s12890-020-01201-y. PMID 32532226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At least 35 patients were planned to be recruited in the study. However, in total, 17 patients entered into the study and completed.
  Reason for termination was challenge with enrollment and recruitment. A significant decrease in the eligible patient population was main driver.
Groups:
- Tobramycin Inhalation Solution(TIS): 300mg nebulized Tobramycin (Tobramycin inhalation solution(TIS)) twice a day (BID) 28days on / 28 days off
- Tobramycin Inhalation Powder (TIP): TOBI Podhaler (Tobramycin inhalation powder(TIP), equivalent dry powder)twice a day (BID) 28days on / 28 days off
Period: Overall Study
Arm/Group | Tobramycin Inhalation Solution(TIS) | Tobramycin Inhalation Powder (TIP)
Started | 5 | 12
Completed | 5 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tobramycin Inhalation Solution(TIS) | Tobramycin Inhalation Powder (TIP) | Total
Number analyzed (Participants) | 5 | 12 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.2 (8.26) | 28.9 (9.79) | 26.4 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 9 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 12 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lung Clearance Index (LCI) After 4 Weeks Following Onset of Study
Description: The Lung Clearance Index (LCI), measured by Multiple Breath Washout of a tracer gas reflects the obstruction of airways in the lung. Wash-out was completed by definition at the time point when the inhaled gas concentration declined to 2.5% of its concentration at baseline. Washout took longer in patients with more severe disease as gas was trapped in narrowed airways (leading to a higher LCI). A LCI of 7.5 and below is normal.
Time Frame: Baseline, week 4
Population: Safety Set consisted of All 17 patients (in both arms: TIS and TIP) that entered the study (provided informed consent) and had been exposed to at least one dose of study drug. The efficacy analysis was based on safety set of Tobramycin ALL and not for each separate dosage form arm.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tobramycin ALL
Number analyzed (Participants) | 17
units on a scale
  Baseline | 17.985 (1.1494)
  Week 4 | 17.101 (0.8409)
Statistical Analysis 1: Comparison: Tobramycin ALL; Test type: Other; p = 0.4099, ANOVA

2. Secondary Outcome: Change From Baseline of Forced Expiratory Volume at 1 Second (FEV1) After 4 Weeks Following Onset of Study
Description: Change of FEV1 (Forced expiry volume in the first second) measured by Spirometry
Time Frame: Baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % predicted
Arm/Group | Tobramycin ALL
Number analyzed (Participants) | 17
% predicted
  Baseline | 76.964 (4.5121)
  Week 4 | 77.481 (4.9877)
Statistical Analysis 1: Comparison: Tobramycin ALL; Test type: Other; p = 0.6961, ANOVA

3. Secondary Outcome: Change From Baseline of Colony-forming Units (CFU) After 4 Weeks Following Onset of Study
Description: Microbacterial density of Pseudomonas aeruginosa in Sputum-Samples in CFU (Colony Forming Units) per gram sputum.
Time Frame: Baseline, week 4
Population: Safety Set consisted of All 17 patients (in both arms: TIS and TIP) that entered the study and had been exposed to at least one dose of study drug. The efficacy analysis was based on safety set of Tobramycin ALL and not for each separate dosage form arm. n is the number of patients of safety set with a non-missing value at the specific time point.
Measure: Least Squares Mean (Standard Error); unit: CFU per gram sputum
Arm/Group | Tobramycin ALL
Number analyzed (Participants) | 17
CFU per gram sputum
  Baseline | 56594.3 (28018.89)
  Week 4: number analyzed (Participants) | 10
  Week 4 | 26113.0 (27280.98)
Statistical Analysis 1: Comparison: Tobramycin ALL; Test type: Other; p = 0.3540, ANOVA

4. Secondary Outcome: Change From Baseline in Lung Clearance Index (LCI) After 1 Week
Description: as for outcome 1
Time Frame: Baseline, week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tobramycin ALL
Number analyzed (Participants) | 17
units on a scale
  Baseline | 17.985 (1.1494)
  Week 1 | 17.506 (1.0002)
Statistical Analysis 1: Comparison: Tobramycin ALL; Test type: Other; p = 0.5910, ANOVA

5. Secondary Outcome: Change of Lung Clearance Index (LCI) Between Week 4 (End of Study Drug Inhalation in the Current Treatment Cycle) and Week 8 (Prior to Start of Study Drug Inhalation in the Following Treatment Cycle)
Description: as for outcome 1
Time Frame: week 4, week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tobramycin ALL
Number analyzed (Participants) | 17
Units on a scale
  Week 4 | 17.101 (0.8409)
  Week 8 | 16.489 (1.1473)
Statistical Analysis 1: Comparison: Tobramycin ALL; Test type: Other; p = 0.4249, ANOVA

6. Secondary Outcome: Change of Forced Expiratory Volume at 1 Second(FEV1) Between Week 4 (End of Study Drug Inhalation in the Current Treatment Cycle) and Week 8 (Prior to Start of Study Drug Inhalation in the Following Treatment Cycle)
Description: Change of FEV1 (Forced expiry volume in the first second) measured by Spirometry
Time Frame: week 4, week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % predicted
Arm/Group | Tobramycin ALL
Number analyzed (Participants) | 17
% predicted
  Week 4 | 77.481 (4.9877)
  Week 8 | 78.705 (5.4782)
Statistical Analysis 1: Comparison: Tobramycin ALL; Test type: Other; p = 0.3963, ANOVA

7. Secondary Outcome: Change of Colony-forming Units (CFU) Between Week 4 (End of Study Drug Inhalation in the Current Treatment Cycle) and Week 8 (Prior to Start of Study Drug Inhalation in the Following Treatment Cycle)
Description: Microbacterial density of Pseudomonas aeruginosa in Sputum-Samples in CFU (Colony Forming Units) per gram sputum.
Time Frame: week 4, week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: CFU per gram sputum
Arm/Group | Tobramycin ALL
Number analyzed (Participants) | 17
CFU per gram sputum
  Week 4: number analyzed (Participants) | 10
  Week 4 | 26113.0 (27280.98)
  Week 8: number analyzed (Participants) | 15
  Week 8 | 56285.0 (28022.28)
Statistical Analysis 1: Comparison: Tobramycin ALL; Test type: Other; p = 0.3502, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment through study completion, an average of 11 weeks.
Description: AE additional description
Arm/Group | Tobramycin Inhalation Solution(TIS) | Tobramycin Inhalation Powder (TIP)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/12
Other Adverse Events (participants affected / at risk) | 2/5 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin Inhalation Solution(TIS) (N=5) | Tobramycin Inhalation Powder (TIP) (N=12)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Forced expiratory volume decreased (Investigations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single- site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-08-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT02248922/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT02248922/SAP_001.pdf